CLINICAL TRIAL: NCT01734395
Title: An Observational, Multi-Center Study to Demonstrate That the Change of Attention Measure is Correlated With the Changes of Caregiver's Burden After Treatment With Galantamine in Patients With Alzheimer's Disease
Brief Title: A Study to Show That the Change of Attention Measure is Correlated With the Changes of Caregiver's Burden After Treatment With Galantamine in Patients With Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100958; GAL-KOR-024 (Other: Janssen Korea, Ltd., Korea); GALALZ4045 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Results first posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Caregiver's Burden in Alzheimer's disease; Galantamine; Razadyne; Reminyl
MeSH Terms: conditions — Alzheimer Disease | interventions — Galantamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Galantamine: Patients will receive galantamine 8 mg/day for the first 4 weeks and the dose of galantamine will be increased up to 24 mg (if tolerable).
  Interventions: Drug: Galantamine

INTERVENTIONS:
Drug: Galantamine — This is an observational study. Galantamine 8 mg/day will be administered for the first 4 weeks and later on the dose will increased up to 24 mg (if tolerable). Galantamine dose will be adjusted according to the investigator's discretion.
  Other Names: Razadyne; Reminyl

SUMMARY:
The purpose of this study is to demonstrate that the change of attention measure is correlated with the changes of caregiver's burden after treatment with galantamine.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), prospective (in which the participants are first identified and then followed forward as time passes), observational (study in which the investigators/ physicians observe the patients and measure their outcomes), multi-center (study conducted at multiple sites) study. The study mainly consists of 2 phases including, the screening phase (14 days before administration of study medication) and treatment phase (16 weeks). In the treatment phase, patients will receive galantamine 8 mg/day for the first 4 weeks and later on the dose will be increased up to 24mg (if tolerable). Safety evaluations will include assessment of adverse events. The total duration of the study will be 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease according to the criteria of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), National Institute of Neurological and Communicative Diseases and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA)
* Measuring standard: K-MMSE is 10 to 24
* Patient with reliable Guardian

Exclusion Criteria:

* Patients with brain tumor, nerve syphilis, meningitis, encephalitis, epilepsy
* Major psychiatric patients such as major depression and schizophrenia
* Patients with treatment-resistant gastric and peptic ulcer
* Patients with clinically serious hepatic, renal, lung, endocrinal or metabolic disease (thyroid, parathyroid, pituitary, renal failure, diabetes mellitus)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Alzheimer's disease
Sampling Method: Non-Probability Sample
Enrollment: 1882 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1,882 participants were recruited to the 84 study centers.
Pre-assignment Details: Out of 1,882 participants, 489 participants violated the inclusion/exclusion criteria and were excluded from the full analysis set (FAS). 1,472 participants completed the study. Total 1,393 participants were included in the FAS population.
Groups:
- Galantamine: Galantamine 8 mg/day for first 4 weeks and the dose will be increased up to 24 mg (if tolerable) for next 12 weeks.
Period: Overall Study
Arm/Group | Galantamine
Started | 1882
Completed | 1472
Not Completed | 410
Not completed — Other | 65
Not completed — Lost to Follow-up | 287
Not completed — Lack of Efficacy | 5
Not completed — Adverse Event | 40
Not completed — Withdrawal by Subject | 10
Not completed — Missing the reasons for not completed | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were determined in Full Analysis Set (FAS) population. Out of 1,882 enrolled participants, 1,393 participants were included in the FAS and 489 participants were excluded due to violation of the inclusion/exclusion criteria.
Arm/Group | Galantamine
Number analyzed (Participants) | 1393
Age Continuous [Mean (Standard Deviation); unit: Years] | 74.11 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 895
  Male | 498
Severity of symptoms of dementia [Number; unit: Participants] — Dementia is a general term for a decline in mental ability severe enough to interfere with daily life. Some of the most common form of dementia is Alzheimer's disease. The severity of dementia is divided as: (1) Suspected dementia (it is also named as Pre-dementia - often mistakenly attributed to ageing or stress), (2) Mild dementia, (3) Moderate dementia, (4) Sever dementia, and (5) Late (very severe) dementia.
  Participants
    Suspected dementia | 27
    Moderate dementia | 668
    Severe dementia | 94
    Late (very severe) dementia | 6
    Mild dementia | 598

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 16 in Attention Questionnaire Scores (AQS)
Description: AQS evaluates the attention of participants with dementia and is designed for their caregivers to evaluate the participant's attention directly. It has 15 questions devised to be suitable for cultural characteristics of Korea through the standardization study considering education and gender/culture gap. Each question is scored from 0 to 2 (0=never, 1=occasionally, 2=usually). In questions 1 to 8, the lower participant attention ability rated the higher score (AQS1), In questions 9 to 15, the higher participant attention ability rated the higher score (AQS2). The total score is calculated by the formula: 16-AQS1+AQS2 and the range is from 0 to 30. Higher score means better attention ability of participant.
Time Frame: Baseline (Week 1 [Day 1]), Week 16
Population: FAS (Full Analysis Set) was used for the analysis. The FAS population was defined as the participants who satisfied the inclusion/exclusion criteria and received the study drug at least once and whose evaluation visit was performed at least once in addition to the visit at baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Galantamine
Number analyzed (Participants) | 1393
Units on a scale | -1.19 (4.56)
Statistical Analysis 1: Comparison: Galantamine; Test type: Superiority or Other; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = -1.19, 95% CI 2-sided [-1.4262 to -0.9467], Standard Deviation 4.56

2. Primary Outcome: Change From Baseline at Week 16 in Burden Interview (BI) Scores
Description: BI is designed to evaluate subjective stress dementia patients' caregivers experience in relation to caregiving. It has total 22 questions with 4 options each and the calculated scores are from 1 to 88 (0-20 = Little or no burden, 21-40 = Mild to moderate burden, 41-60 = Moderate to severe burden, 61-88 = Severe burden). Higher scores indicate worsening.
Time Frame: Baseline, Week 16
Population: FAS was used for the analysis. The FAS population was defined as the participants who satisfied the inclusion/exclusion criteria and received the study drug at least once and whose evaluation visit was performed at least once in addition to the visit at baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Galantamine
Number analyzed (Participants) | 1393
Units on a scale | 1.48 (10.69)
Statistical Analysis 1: Comparison: Galantamine; Test type: Superiority or Other; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = 1.48, 95% CI 2-sided [0.9188 to 2.0438], Standard Deviation 10.69

3. Secondary Outcome: Change From Screening at Week 16 in Mini Mental State Exam Scores (MMSE)
Description: MMSC is a brief 30-point questionnaire test that is used for the assessment of dementia patients' cognitive impairment. Evaluation of points are as: 24-30 = No cognitive impairment, 18-23 = Mild cognitive impairment, 0-17 = Severe cognitive impairment. Lower scores indicate worsening.
Time Frame: Baseline, Week 16
Population: FAS was used for the analysis. The FAS population was defined as the participants who satisfied the inclusion/exclusion criteria
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Galantamine
Number analyzed (Participants) | 1393
Units on a scale | -0.69 (2.43)
Statistical Analysis 1: Comparison: Galantamine; Test type: Superiority or Other; p < .0001, t-test, 2 sided; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-0.814 to -0.5586], Standard Deviation 2.43

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Description: Participants who received the study drug at least once were analysed. There was 9 serious adverse events in 7 participants were reported and no other adverse event in more than 5% of participants were reported.
Arm/Group | Galantamine
Serious Adverse Events (participants affected / at risk) | 7/1882
Other Adverse Events (participants affected / at risk) | 0/1882
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galantamine (N=1882)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Asthenia (General disorders) | 2 (2)
Death (General disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days